CLINICAL TRIAL: NCT03485755
Title: The Evolution of the Skin Microbiome of Children Approximately Ages 8-10 Years of Age
Brief Title: Pediatric Microbiome Study With Children Now Approximately 8-10 Years Old.
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Other Study IDs: CCSSKA000104
Record Dates: First submitted 2018-03-08; First posted 2018-04-02 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
Keywords: microflora; microbiome; bacteria taxa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Children 8-10 years of age
- Biological Mothers: Biological mothers of children now ages 8-10 years of age

SUMMARY:
Single site study involving Biological Mothers and their children approximately 8-10 years old to assess the predominant microflora and skin physiology.

ELIGIBILITY:
Inclusion Criteria:

* Must be the biological mother of a child (approximately age 8-10 years) enrolled in the study
* All subjects are to have normal healthy skin and no presence of pre-existing or dormant dermatologic skin conditions;
* Willing to use only the provided cleansing product during the washout time period;
* Willing to refrain from topical product use on the skin for the duration of the study. Topical products that should not be used include moisturizers, lotions, sunscreens, oils, tanners;
* Willing to refrain from swimming, using hot tubs, excessive sun exposure or tanning beds during the course of this study;

Exclusion Criteria:

* Presents with a skin condition that may influence the outcome of the study (specifically psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, active skin cancer) a

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and their biological mothers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Microbial Community Diversity for Children | Day 1
  Swabs will be collected from the volar forearm, forehead and cheek for analysis based on the Shannon Index

SECONDARY OUTCOMES:
Microbial Community Diversity for Adults | Day 1
  swabs will be collected from the volar forearm, forehead and cheek for analysis based on the Shannon Index
Microbial Community Richness for Children | Day 1
  swabs will be collected from the skin for analysis to determine the total number of different bacterial taxa detected
Microbial Community Richness for Adults | Day 1
  swabs will be collected from the volar forearm, forehead and cheek for analysis to determine the total number of different bacterial taxa detected
Skin Barrier Function | Day 1
  Trans Epidermal Water Loss (TEWL) will be used to assess the skin barrier function
Skin pH | Day 1
  skin pH will be assessed by pH meter

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L Moskovitz, MD, Principal Investigator — Bruce L Moskovitz MD - private consultant
Locations (1):
- Consumer Experience Center, Skillman, New Jersey, United States

REFERENCES:
- See also: Redacted Clinical Study Report — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSSKA000104&attachmentIdentifier=8f7ee7fb-3df4-4ce7-9abf-8dffe2a67754&fileName=Ped_Microbiome___CCSSKA000104___Redacted_CSR.pdf&versionIdentifier=